CLINICAL TRIAL: NCT00796315
Title: A Single-dose, Open-label, Multi-center Study Evaluating the Pharmacokinetics of Doxylamine Succinate in Children Ages 2 to < 18 Years
Brief Title: Study Evaluating the Pharmacokinetics of Doxylamine Succinate in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Collaborators: Consumer Healthcare Products Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2008014
Record Dates: First submitted 2008-11-18; First posted 2008-11-24 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Allergic Rhinitis; Upper Respiratory Infection
Keywords: Pharmacokinetic study
MeSH Terms: conditions — Rhinitis, Allergic; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxylamine Succinate (USP) (Experimental): Doxylamine Succinate United States Pharmacopeia (USP)
  Interventions: Drug: Doxylamine Succinate USP

INTERVENTIONS:
Drug: Doxylamine Succinate USP — One dose of liquid, dosing range 3.125mg/7.5mL - 12.5mg/30mL
  Other Names: Doxylamine Succinate United States Pharmacopeia (USP)

SUMMARY:
The primary goal of this study is to characterize the pharmacokinetics of doxylamine succinate in children ages 2 to < 18 years. Once characterized, these pediatric pharmacokinetic data will be pooled with historical adult PK data from other studies to assess whether the existing Over-the-Counter (OTC)doses provide comparable systemic drug exposure as that associated with efficacy in adults.

ELIGIBILITY:
Inclusion Criteria:

* are male or female children ages 2 to < 18 years, with a minimum weight of 24 lbs and > 5th percentile and < 95th percentile for weight based on age and sex, at the time of dosing study medication
* had a previous diagnosis of allergic rhinitis, or had a history of frequent upper respiratory infections (URI)/common cold and either be symptomatic, or at risk for future URI, including each of the following 3 criteria

  * Frequency Criterion: > 6 infections per year for children aged 2 to <6 years of age and > 4 infections per year for children aged 6 to < 18 years of age
  * Crowding Criterion: 4 persons living in the home or 3 persons sleeping in one bedroom
  * Exposure Criterion: another family member in the home who is ill with URI / common cold or a child in the family who is attending preschool or school with 6 children in the group.
* are in good general health
* are likely to be compliant and complete the study and have parent(s) or legally authorized representative(s) likely to be compliant and complete the study according to the Investigator
* whose parent(s) or legally authorized representative(s) have signed and dated an Institutional Review Board (IRB)-approved consent form for the subject to participate in the study
* must have signed an assent form as required by the site's IRB
* if post-menarchal females, subjects must have a negative urine pregnancy test at screening and check-in, or serum pregnancy test at screening, if site required;
* if post-menarchal females, subjects must practice abstinence or use an effective form of birth control (eg, intrauterine device, low dose oral contraceptives [ 50g ethinyl estradiol], contraceptive implants or injections, diaphragm with spermicide, cervical cap, or consort use of condom) for at least 3 months before being enrolled in the study.

Exclusion Criteria:

* has any history or presence of the following medical conditions: peptic ulcer, pyloroduodenal obstruction or other gastrointestinal disease; renal or hepatic disease; diabetes mellitus; hyperthyroidism; cardiovascular disease;increased ocular pressure or glaucoma; endocrine, metabolic, hematologic or neoplastic disease; seizure disorder; chronic respiratory diseases including asthma, emphysema and chronic bronchitis; autoimmune disease; immunodeficiency tuberculosis; bladder neck obstruction; significant dermatologic condition.
* has a known sensitivity or allergy to doxylamine succinate
* has a history of a severe allergic reaction to any drug or has multiple food/drug allergies
* experienced febrile illness greater than 100°F within 7 days prior to dosing
* reports any known enzyme-inducer, enzyme-inhibitor, or reported chronic exposure to enzyme-inducers such as paint solvents or pesticides within 30 days prior to dosing, unless approved by the Sponsor
* reports any other prescription drug or herbal remedy usage within 14 days prior to dosing except for low dose contraceptives, unless approved by the Sponsor
* reports any non-prescription drug or supplemental vitamin usage within 5 days prior to dosing
* unwillingness to refrain from caffeine or other xanthine-containing beverages, including coffee and tea, alcohol, grapefruit juice, chocolate, or Seville oranges 24 hours prior to admission and throughout the study
* reported use of tobacco, smoking cessation products, or products containing nicotine within 3 months prior to Screening
* has an acute illness (except as described in Section 3.3.1 Inclusion Criterion b) within 14 days prior to dosing; unless approved by the Sponsor;
* has any laboratory value outside the laboratory reference range considered clinically significant by the Investigator
* has a history or diagnosis of Hepatitis B, Hepatitis C, human immunodeficiency virus (HIV), or thyroid disease
* has a history of alcohol or illicit drug use or a positive urine drug of abuse screen
* are pregnant or lactating (post-menarchal female subjects should be made aware that pregnancy testing will occur during the study, and that if they are sexually active they must take appropriate steps to ensure they do not become pregnant during the study)
* has made a blood donation or plasma donation within 4 weeks prior to dosing;
* has participated in another investigational drug study protocol within 30 days prior to dosing (Day -1)
* has a history or presence, upon clinical evaluation, of any illness or condition that might impact safety of the subject with test product administration or evaluability of drug effect, based on the Investigator's discretion
* is unable to avoid driving, operating machinery, or other tasks that require alertness during the study.
* is unable or unwilling to avoid contact sports, strenuous exercises (e.g. weight lifting), exercises for which they are not trained or conditioned or intramuscular injection for at least 1 week before baseline visit when creatine phosphokinase (CPK) will be evaluated

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molly Seeck, BS, JD, Study Director — Procter and Gamble
Locations (6):
- United States (6):
  - Dana Best, MD, Washington D.C., District of Columbia
  - Janice E. Sullivan, MD, Louisville, Kentucky
  - Margaret Ann Springer, MD, Shreveport, Louisiana
  - Bridgette Jones, MD, Kansas City, Missouri
  - Alex Kemper, Pharm D, Durham, North Carolina
  - Jeffrey L Blumer, MD, PhD, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow is described by three different age groups based on dosing differences for each group
Groups:
- Subjects Aged 2-5 Years (Doxylamine Succinate): Ages 2-5 years. Doxylamine Succinate USP : One dose of liquid, dosing range 3.125mg/7.5mL - 12.5mg/30mL.
- Aged 6-11 Years (Doxylamine Succinate: Ages 6-11 years. Doxylamine Succinate USP : One dose of liquid, dosing range 3.125mg/7.5mL - 12.5mg/30mL.
  Note: One subject (age group 6-11) was unable to meet protocol criteria (spit out a portion of his dosage) and was discontinued.
- Subjects Aged 12-17 Years (Doxylamine Suc: Ages 12-17 years. Doxylamine Succinate USP : One dose of liquid, dosing range 3.125mg/7.5mL - 12.5mg/30mL.
Period: Overall Study
Arm/Group | Subjects Aged 2-5 Years (Doxylamine Succinate) | Aged 6-11 Years (Doxylamine Succinate | Subjects Aged 12-17 Years (Doxylamine Suc
Started | 9 | 17 | 15
Completed | 9 | 16 | 15
Not Completed | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Doxylamine Succinate USP: Doxylamine Succinate, United States Pharmacopeia (USP): One dose of liquid, dosing range 3.125mg/7.5mL - 12.5mg/30mL.
Arm/Group | Doxylamine Succinate USP
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years]
  Subjects Aged 2-5 years | 3.6 (1.1)
  Subjects Aged 6-11 years | 8.5 (1.5)
  Subjects Aged 12-17 years | 14.5 (1.8)
Sex/Gender, Customized [Number; unit: participants]
  Male, Ages 2-5 | 7
  Female, Ages 2-5 | 2
  Male, Ages 6-11 | 9
  Female, Ages 6-11 | 8
  Male, Ages 12-17 | 9
  Female, Ages 12-17 | 6
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: AUC of Doxylamine
Description: Area under the time-concentration curve for Doxylamine from 0 to 72 hours post-dose plus an extrapolated area from 72 hours to infinity.
Time Frame: 72 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Subjects Aged 2-5 Years: Ages 2-5 years. Subjects received a dose of either 3.125 or 4.17 mg Doxylamine Succinate USP (exact dose dependent upon body weight)
- Subjects Aged 6-11 Years: Ages 6-11 years. Subjects received a dose of 4.17 or 6.25 or 8.33 or 10.42 mg Doxylamine Succinate USP (exact dose dependent upon body weight). Note: One subject (age group 6-11) was unable to meet protocol criteria (spit out a portion of his dosage) and was discontinued.
- Subjects Aged 12-17 Years: Ages 12-17 years. All subjects received a dose of 12.5 mg Doxylamine Succinate USP
Arm/Group | Subjects Aged 2-5 Years | Subjects Aged 6-11 Years | Subjects Aged 12-17 Years
Number analyzed (Participants) | 9 | 16 | 15
ng*h/mL | 461.9 (51.2) | 810.1 (27.9) | 827.0 (45.4)

2. Primary Outcome: Cmax of Doxylamine
Description: Maximum concentration of Doxylamine from 0 to 72 hours post-dose
Time Frame: 72 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Subjects Aged 2-5 Years: Ages 2-5 years. Doxylamine Succinate USP
- Subjects Aged 6-11 Years: Ages 6-11 years. Doxylamine Succinate USP
- Subjects Aged 12-17 Years: Ages 12-17 years. Doxylamine Succinate USP
Arm/Group | Subjects Aged 2-5 Years | Subjects Aged 6-11 Years | Subjects Aged 12-17 Years
Number analyzed (Participants) | 9 | 16 | 15
ng/mL | 50.1 (22.5) | 65.8 (19.9) | 63.2 (42.9)

ADVERSE EVENTS:
Time Frame: Adverse Events collected until discharge from study, approximately 72 hours after dose
Groups:
- Aged 6-11 Years: Ages 6-11 years. Doxylamine Succinate USP
Arm/Group | Subjects Aged 2-5 Years | Aged 6-11 Years | Subjects Aged 12-17 Years
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 5/9 | 4/17 | 7/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Aged 2-5 Years (N=9) | Aged 6-11 Years (N=17) | Subjects Aged 12-17 Years (N=15)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 4 (5) | 3 (3) | 5 (5)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Incidences of mild sedation are consistent with doxylamine's indication as an OTC sleep aid. Conclusive evaluation of sedation couldn't be undertaken in the absence of a control group. Also, children may nap in daytime confounding sedation assessment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator and Sub-Investigators agree that all data, calculations, interpretations, opinions, and recommendations regarding the study will be the property of the Sponsor. The Investigator agrees to consider the results as information subject to confidentiality and use restrictions.